CLINICAL TRIAL: NCT04428710
Title: Cancer Genetic Counseling and Emotional Response in Spanish Population
Brief Title: Assessment Psychological Distress for Cancer Heredity Test
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Gemma Costa Requena, PhD Clinical psychologist, Hospital Universitario La Fe
Other Study IDs: Cancer Genetic Counseling.PSI
Record Dates: First submitted 2020-05-30; First posted 2020-06-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Cancer; Psychological Distress; Hereditary Diseases; Genetic Counseling
MeSH Terms: conditions — Neoplasms; Genetic Diseases, Inborn | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted to cancer genetic counseling test: Participants were recruited from all consecutive patients referred to the Cancer Genetic Program at the Hospital Universitari i Politècnic la Fe.
  Interventions: Other: assessment with psychometric questionnaire

INTERVENTIONS:
Other: assessment with psychometric questionnaire — At the initial genetic consultation patients are informed about hereditary cancer risk and the genetic testing process. At the second genetic counseling appointment, after patients done tests, all participants were informed about the study purpose, and they signed the informed consent before the psychometric assessment. Those patients who agreed to participate, they were given the questionnaires to fill in. Also, background characteristics were reported including age, marital relationship, level of education, psychiatric antecedents.
  The time for completion the self-report measures was about 10 minutes. The psychometric assessment was occurred prior to delivering the results of genetic testing.

SUMMARY:
The study of hereditary cancer related syndromes allows reducing the risk of suffering in cancer to patients and close relatives. The objective of this study will be to evaluate the prevelance of psychological morbidity in patients attended at cancer genetic counselling unit, and to determine the socio-demographic and clinical factors that influence it.

A descriptive cross-sectional study will be carried out. Patients attented at the cancer genetic counselling unit, who have criteria for conducting a genetic syndrome test related to hererditary cancer, will be consecutively evaluated.

To knowing the psychological morbidity it is relevant to providing care for these patients.

DETAILED DESCRIPTION:
Nowadays several familial cancer syndromes that confer a high lifetime risk of cancer can be identified with genetic testing. The psychological impact of genetic testing and the rates of psychological distress in patients undergoing genetic testing vary between 6 to 65% depending on socio-demographic or clinical characteristics.

The effect of baseline distress on post-testing assessments tended to decrease or show little change over time, it may be important to target patients with high baseline distress for additional counseling or intervention both pre-testing and over time.The most robust predictor of future distress is baseline distress, additional factors were associated with cancer risk perception considering family history of cancer, patient's affected or unaffected with cancer, etc...

It is relevant to developing and providing care for these patients, it has been demonstrated that enhanced genetic counseling with clinical psychologist to facilitate decision-making process, managing family concerns promoting their communication with and involvement of family members, and attending their emotional distress, can be beneficial. Also, cancer genetic counseling may promote patient use of personal resources and enhance patient health literacy about their syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Factors presumed predictive for hereditary cáncer
* They agreed to participate in the research.

Exclusion Criteria:

* Patients with cognitive impairment
* Patients with difficulties to read and understand Spanish language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from all consecutive patients referred to the Cancer Genetic Program at the Hospital Universitari i Politècnic la Fe.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To determinate the prevalence of psychological distress of patients studied of the different hereditary cancer syndromes attended at Cancer Genetic Counseling Unit | Data collection for two years
  The Hospital Anxiety and Depression Scale (HADS), it is consisting of two subscales with seven items respectively, anxiety (HADS-A) and depression (HADS-D) symptomatology. The questionnaire is used to evaluate psychological distress in non-psychiatric settings. In general medical outpatients the optimal cut-off point for the screening for psychiatric morbidity seems to be 12, for screening depressive symptomatology seems to be 5 score and 8 (range 7-10) for screening anxiety symptomatology. In Spanish population the HADS demonstrated a good internal consistency and optimal psychometric properties.
To determinate cáncer worry of patients studied of the different hereditary cancer syndromes attended at Cancer Genetic Counseling Unit | Data collection for two years
  Cancer Worry Scale. (CWS), consists of the six-item scale measures concerns about developing cancer, and the impact of these concerns on performing daily tasks among patients at risk for hereditary cancer. The questionnaire are rated on a 4-point Likert scale ranging from "never" to "almost always", with a total value ranging from 6 (minimal worry) to 24 (maximum worry). CWS presented good reliability coefficient in Spanish samples at risk for hereditary cancer.
To determinate the prevalence of psychological morbidity of patients studied of the different hereditary cancer syndromes attended at Cancer Genetic Counseling Unit | Data collection for two years
  The General Health Questionnaire (GHQ-28), measures psychological distress, which is consisting of social functioning, somatic symptoms, anxiety/sleep disturbances, and depression. Each item was scored from 0 to 3. Higher scores indicating greater psychological morbidity, with a cutting score of 5/6 to identify psychiatric morbidity. The Spanish version of the GHQ-28 had adequate psychometric properties.

SECONDARY OUTCOMES:
Find out differences on psychological distress regarding the hereditary syndrome studied at the cancer genetic counseling. | Data collection for two years
  Psychometric questionnaire. Hospital Anxiety and Depresion Scale (HADS) , it is consisting of two subscales with seven items respectively, anxiety (HADS-A) and depression (HADS-D) symptomatology. The questionnaire is used to evaluate psychological distress in non-psychiatric settings. The optimal cut-off point for screening psychiatric morbidity seems to be 12, for screening depressive symptomatology seems to be 5 score and 8 (range 7-10) score for screening anxiety symptomatology. In Spanish population the HADS demonstrated a good internal consistency and optimal psychometric properties.
Identify differences in cancer worry regarding the hereditary syndrome studied at the cancer genetic counseling. | Data collection for two years
  Cancer Worry Scale (CWS). this questionnaire consists of the six-item measures concerns about developing cancer and the impact of these concerns on performing daily tasks among patients at risk for hereditary cancer. The questionnaire are rated on a 4-point Likert scale ranging from "never" to "almost always", with a total value ranging from 6 (minimal worry) to 24 (maximum worry). CWS presented good reliability coefficient in Spanish samples at risk for hereditary cancer.
Psychometric analysis of the questionnaires used to assess psychological distress and cancer worry | Data collection for two years
  Impact of Event Scale (IES), is a self-report measure for distress in relation to a stressful life event, which in our study is cancer risk. IES is using 15 items to measures psychological distress on two subscaless, with intrusion (the extent to which patients are overwhelmed by thoughts and feelings about cancer) and avoidance (tendency to avoid thoughts and feelings about cancer). The intrusion subscale has seven items, the avoidance subscale eight items. Each item is scored from 0 to 5. The psychometric properties of IES are good in samples with increased risk for hereditary breast cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Costa-Requena G, Garcia-Garijo M, Richart-Aznar P, Segura-Huerta A. Comparison of psychological distress for breast, ovarian and colorectal cancer predisposition in a Spanish sample at high risk of hereditary cancer. Eur J Cancer Prev. 2022 Sep 1;31(5):482-486. doi: 10.1097/CEJ.0000000000000734. Epub 2021 Dec 15. PMID 36165038
- [Derived] Costa-Requena G, Garcia-Garijo M, Richart-Aznar P, Segura-Huerta A. Psychiatric symptoms in a Spanish sample with hereditary cancer risk. J Community Genet. 2022 Jun;13(3):339-346. doi: 10.1007/s12687-022-00580-5. Epub 2022 Feb 8. PMID 35133604